CLINICAL TRIAL: NCT06931054
Title: Combination of Acupuncture, Auricular Acupressure and Nicotine Replacement Therapy for Smoking Cessation: A Randomized Controlled Trial
Brief Title: Combination of Acupuncture, Auricular Acupressure and Nicotine Replacement Therapy for Smoking Cessation
Acronym: acupuncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acupuncture_protocol_v3; 23B2/056A_R1 (Other Grant/Funding Number: Chinese Medicine Development Fund)
Record Dates: First submitted 2025-04-14; First posted 2025-04-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Smoking
Keywords: Acupuncture; Smoking cesastion; NRT; Acupressure
MeSH Terms: conditions — Smoking | interventions — Acupuncture Therapy; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Acupuncture, auricular acupressure, nicotine replacement therapy and smoking cessation counseling
  Interventions: Other: Acupuncture; Drug: Nicotine Replacement therapy; Behavioral: Smoking cessation counseling; Other: Auricular acupressure
- Control group 1 (Sham Comparator): Sham acupuncture, sham acupressure, nicotine replacement therapy and smoking cessation counseling
  Interventions: Drug: Nicotine Replacement therapy; Behavioral: Smoking cessation counseling; Other: Sham acupressure; Other: Sham acupuncture
- Control group 2 (Active Comparator): Nicotine replacement therapy, smoking cessation counseling
  Interventions: Drug: Nicotine Replacement therapy; Behavioral: Smoking cessation counseling

INTERVENTIONS:
Other: Acupuncture — The principle of traditional acupuncture and auricular acupressure is to alleviate withdrawal symptoms. Acupuncture therapy for smoking cessation is generally considered safe, but some people may experience mild side effects. These can include soreness, bruising, or bleeding at the needle insertion sites, dizziness, fatigue, or lightheadedness after treatment. Occasionally, individuals may feel nausea or discomfort during or after the session. In rare cases, infections can occur if proper hygiene protocols are not followed. Overall, most side effects are temporary and resolve shortly after treatment.
  Primary Acupoints The selection of body acupuncture points follows specific guidelines[11-12], including three head points (Baihui, Shenting, Yintang ), three hand points (Neiguan, Kongzui, Lieque), and three foot points (Zusanli, Sanyinjiao, Taichong). For auricular acupoints, selection is based on corresponding areas (Mouth), syndrome differentiation of zang-fu organs and meridians (Hea
  Arms: Experimental group
Drug: Nicotine Replacement therapy — Each eligible participant will be prescribed a two-week supply of NRT by a registered smoking cessation nurse following the initial counseling session. The nurse will determine the appropriate type and dosage of NRT based on the participant's level of nicotine dependence and lifestyle habits, and provide instructions on how to use the medication. NRT can cause some potential side effects such as nausea, headaches, dizziness, and insomnia, with vivid dreams being common for those using patches. Method-specific side effects include skin irritation from patches, mouth or throat irritation from gums or lozenges, and nasal or throat discomfort from inhalers and sprays. These symptoms usually lessen as the body adjusts, but persistent or worsening side effects may require medical attention. According to current smoking cessation medication guidelines from the Department of Health[10], participants who smoke 20 or more cigarettes per day will be prescribed 4 mg nicotine gum (or lozenges) or 2
Behavioral: Smoking cessation counseling — The first step for smoking cessation nurses is to assess each participant's smoking behavior using a baseline questionnaire. In the second step, informed consent will be obtained from the participants. The third step involves smoking cessation counseling using the 5A (Ask, Advise, Assess, Assist, Arrange) and 5R (Relevance, Risks, Rewards, Roadblocks, Repetition) frameworks as outlined in the smoking cessation manual published by the Department of Health. During this step, the nurse will also assess the type and dosage of NRT suitable for the participant. In the fourth step, participants will be introduced to TCM therapies, and arrangements will be made for consultations with a TCM practitioner.
Other: Auricular acupressure — First, one ear will be routinely disinfected with 75% medical ethanol. In the experimental group, the auricular acupressure tape contains Semen Vaccariae. Using forceps or tweezers, an auricular acupressure tape will be applied to specific acupoints on one ear for participants in the experimental group, followed by pressing the tape for 1 minute. The auricular tape will remain in place for two days, and participants will be instructed to self-press the acupoints 3 to 5 times daily, for 1 minute per acupoint each time. During the use of the auricular acupressure, if withdrawal symptoms occur, participants can immediately press the acupoints. The pressure applied should be tolerable, and the pressing duration should last until the withdrawal symptoms subside. Participants will also record the number of presses each day.
  Arms: Experimental group
Other: Sham acupressure — The sham tape resembles the genuine auricular acupressure tape with Semen Vaccariae but is a regular adhesive tape designed to minimize stimulation of the acupoints.
  The sham auricular tape will be applied to non-smoking cessation acupoints, including:
  * Elbow Acupoint located in the third section of the triangular fossa between the middle cartilage and the rim cartilage of the ear, primarily used for treating elbow pain.
  * Ankle Acupoint located near the apex of the superior crus of the antihelix, used for treating arthritis.
  * Urethra Acupoint located on the helix above the rectum acupoint, used for treating symptoms such as frequent urination or painful urination.
  Arms: Control group 1
Other: Sham acupuncture — The TCM practitioner will perform needle insertion 2-3 mm beside the selected acupoints (at non-specific "sham" points) using normal needling techniques but without manipulating the needles, in order to minimize any physiological effects.
  Arms: Control group 1

SUMMARY:
The aims of this study include: (1) to evaluate whether a combined smoking cessation treatment of acupuncture, auricular acupressure, and nicotine replacement therapy (NRT) is more effective in improving smoking cessation rates at a 6-month follow-up compared to NRT alone; (2) to assess whether the combined smoking cessation treatment of acupuncture, auricular acupressure, and NRT increases the incidence of side effects compared to NRT alone; (3) to evaluate whether the combined smoking cessation treatment of acupuncture, auricular acupressure, and NRT is more effective in reducing withdrawal symptoms compared to NRT alone. This study will randomly assign participants into three groups. The total sample size is set at 270 participants, with each group consisting of 90 participants. The randomization ratio is 1:1:1.

DETAILED DESCRIPTION:
The aims of this study include: (1) to evaluate whether a combined smoking cessation treatment of acupuncture, auricular acupressure, and nicotine replacement therapy (NRT) is more effective in improving smoking cessation rates at a 6-month follow-up compared to NRT alone; (2) to assess whether the combined smoking cessation treatment of acupuncture, auricular acupressure, and NRT increases the incidence of side effects compared to NRT alone; (3) to evaluate whether the combined smoking cessation treatment of acupuncture, auricular acupressure, and NRT is more effective in reducing withdrawal symptoms compared to NRT alone. This study will randomly assign participants into three groups. The total sample size is set at 270 participants, with each group consisting of 90 participants. The randomization ratio is 1:1:1.

The intervention group will receive a combination of acupuncture, auricular acupressure, and NRT as a smoking cessation treatment. Control Group 1 will receive a sham version of the combined treatment (i.e., retractable needles that do not penetrate the skin and placebo auricular acupressure). Neither the participants in the experimental group nor those in Control Group 1 will know their group assignment, ensuring a double-blind, 3-arm RCT. Control Group 2 will receive NRT and undergo a standard Chinese medicine general consultation (including observation, auscultation and olfaction, inquiry, pulse-taking, and general health advice) during the initial visit, but will not receive acupuncture or auricular acupressure. Participants in the experimental group and Control Group 1 will not be aware of their specific group assignment. The study protocol will follow the CONSORT guidelines and will seek approval from the university's research ethics committee. Smoking cessation nurses or counsellors will deliver the counseling, The 8-week and 26-week follow up outcome assessments will be done by research assistants and should be blinded of group allocation. Self-reported quitters at 26-week follow-up will be invited for a biochemical validation.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 or older.
2. Individuals who consume at least 10 traditional cigarettes per day.
3. Individuals with access to a smartphone for communication and internet use.
4. Individuals who are able to read and write Chinese.

Exclusion Criteria:

1. Previous use of acupuncture for smoking cessation or any other condition.
2. Skin problems related to diabetes.
3. Hyperthyroidism.
4. Hospitalized at Intensive Care Unit in the past 4 weeks.
5. Severe cardiovascular diseases.
6. Pregnancy.
7. Breastfeeding.
8. History of severe adverse reactions to acupuncture.
9. Current use of blood-thinning medication or having a bleeding disorder.
10. Current use of other smoking cessation services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical validated tobacco abstinence at 26-week follow-up | 26-week follow-up
  Biochemically verified quitting is defined as a carbon monoxide (CO) level in exhaled breath measured by a CO monitor of less than or equal to 3 ppm, and a salivary cotinine level of less than or equal to 30 ng/ml, as tested by a cotinine test strip.

SECONDARY OUTCOMES:
Biochemical validated tobacco abstinence at 8-week follow-up | 8-week follow-up
  Biochemically verified quitting is defined as a carbon monoxide (CO) level in exhaled breath measured by a CO monitor of less than or equal to 3 ppm
Self-reported 7-day point prevalence abstinence at 8-week follow-up | 8-week follow-up
  Self-reported 7-day point prevalence abstinence
Self-reported 7-day point prevalence abstinence at 26-week follow-up | 26-week follow-up
  Self-reported 7-day point prevalence abstinence
Incidence rate of side effects/adverse events | 8-week follow-up
  Incidence rate of side effects/adverse events (e.g., needle fainting, bleeding, etc.).
Number of cigarettes smoked per day at the 8-week follow-up | 8 weeks
  Number of cigarettes smoked per day (in smokers)
Number of cigarettes smoked per day at the 26-week follow-up | 26-week follow-up
  Number of cigarettes smoked per day (in smokers)
Withdrawal symptoms | 8 weeks
  Minnesota Nicotine Withdrawal Scale (MNWS), measured through ecological momentary assessment, scale range from 7 to 35, higher scores mean more frequent withdrawal symptoms
Questionnaire of Smoking Urges-Brief (QSU-B) | 8 weeks
  The 10-item Questionnaire of Smoking Urges-Brief (QSU-B) is used to measure the desire and anticipation of smoking

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The participant data can be made available upon requests with justification on legitimite research purposes.

REFERENCES:
- [Background] Shiffman S. Conceptualizing analyses of ecological momentary assessment data. Nicotine Tob Res. 2014 May;16 Suppl 2(Suppl 2):S76-87. doi: 10.1093/ntr/ntt195. Epub 2013 Dec 9. PMID 24323571
- [Background] Clavel F, Benhamou S, Company-Huertas A, Flamant R. Helping people to stop smoking: randomised comparison of groups being treated with acupuncture and nicotine gum with control group. Br Med J (Clin Res Ed). 1985 Nov 30;291(6508):1538-9. doi: 10.1136/bmj.291.6508.1538. No abstract available. PMID 3933739